CLINICAL TRIAL: NCT01539122
Title: A Multi-Centre, Randomized Controlled Study on the Zimmer TM Glenoid Component Compared to Cemented Glenoid Component
Brief Title: Clinical Experience With the Zimmer Trabecular Metal (TM) Glenoid in Total Shoulder Arthroplasty
Acronym: TMGlenoid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Preservation Centre of BC (Other)
Responsible Party: Principal Investigator, Patrick Chin, Principal Investigator, Joint Preservation Centre of BC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMGlenoid H12-00323
Record Dates: First submitted 2012-02-13; First posted 2012-02-27 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: osteoarthritis; shoulder replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TM Glenoid (Active Comparator): Zimmer TM glenoid shoulder replacement component will be used for the glenoid component of the total shoulder replacement.
  Interventions: Device: Zimmer TM Glenoid
- Cemented Glenoid (Active Comparator): Cemented glenoid shoulder replacement component
  Interventions: Device: Cemented Glenoid

INTERVENTIONS:
Device: Zimmer TM Glenoid — The Zimmer TM glenoid will be used for the glenoid shoulder replacement component.
  Other Names: Zimmer Trabecular Metal Glenoid
  Arms: TM Glenoid
Device: Cemented Glenoid — A cemented glenoid will be used for the glenoid component of the total shoulder replacement.
  Other Names: Cemented all-polyethylene glenoid component (Zimmer)
  Arms: Cemented Glenoid

SUMMARY:
The objective of this randomized controlled study is to obtain outcomes data on the Zimmer TM glenoid component by analysis of standard scoring systems and radiographs in comparison to the cemented glenoid component. In addition, the investigators plan to provide cost analysis based on the economic data collected to justify the cost difference between both implants.

Patients with acceptable glenoid bone stock will be randomized into two groups to be treated with either a TM Glenoid or cemented glenoid component with minimum 2 years follow-up; maximum 10 years follow-up.

Hypothesis: The early and long-term clinical outcomes and radiographic analysis of the TM glenoid components are superior to the cemented glenoid components in total shoulder arthroplasty patients.

DETAILED DESCRIPTION:
Total shoulder arthroplasty is successful in relieving pain and restoring function to the joint, but chronic loosening of the glenoid implant remains a common complication. The Zimmer Trabecular Metal (TM) Glenoid is a monoblock implant for reconstructive total shoulder arthroplasty. To date, no published clinical data is available to confirm evidence on the effectiveness of this specific product.

The purpose of this prospective study is to obtain both short and long-term clinical outcomes data on the Zimmer TM Glenoid by analysis of standard scoring systems and radiographic analysis. The TM Glenoid Component is intended to function within Zimmer, Inc.'s Bigliani/Flatow (B/F) Complete Shoulder Solution. The device is a monoblock glenoid component comprised of a Trabecular Metal base, and is designed to interface and articulate with Zimmer, Inc.'s B/F humeral components. The Trabecular Metal Glenoid is designed with an articular surface that is manufactured from ultra-high molecular weight polyethylene (UHMWPE). The base of the implant has a cruciate TM keel that provides stability and initial fixation using a press-fit between the implant and the bone. Long-term fixation is provided by biological ingrowth into the TM material. Surgical fixation of the trabecular metal device will be obtained via press-fit. Surgical fixation of the comparison all-polyethylene glenoid component will be with Palacos/CoPal bone cement

This is a multi-centre, randomized controlled study to evaluate the clinical and radiological performance of the TM Glenoid in a series of patients with adequate glenoid bone stock receiving a total shoulder replacement. The comparison group will be a consecutive series of randomized patients with implanted cemented all-polyethylene glenoid component. This study will be descriptive in nature and seeks to demonstrate the superiority (or non-inferiority) of the TM Glenoid over cemented all-polyethylene glenoid components.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years minimum and 80 years of age maximum.
* Gender - male and female.
* Primary Diagnosis: Primary Glenohumeral Osteoarthritis
* Informed Consent - patient has signed a 'Patient Informed Consent form'
* Surgery date: Beginning on January 1, 2012
* KEY Inclusion Criteria: The critical inclusion criteria for patient selection for TM or Cemented glenoid prosthesis are based on adequacy of glenoid bone stock/quality at time of implantation. Pre-operative CT scans and intra-operative decision of the surgeon at time of surgery will determine the issue of bone stock/quality.

Exclusion Criteria:

* Age > 80 years
* Significant Bone Loss (classified as concentric vs eccentric; contained vs uncontained) on pre-operative CT scan requiring cemented prosthesis.
* Evidence of major joint trauma, infection, avascular necrosis, cuff tear arthropathy, inflammatory arthropathy, chronic dislocation, massive rotator cuff tear or previous shoulder surgery (other than arthroscopic debridement)
* Preoperative computed tomography scans of the shoulder that showed insufficient glenoid bone stock to allow for implantation of a glenoid prosthesis
* Active joint or systematic infection, significant muscle paralysis, or Charcot arthropathy
* Life expectancy of less than 2 years or unacceptably high operative risk
* Inability to speak or read English
* Psychiatric illness or cognitive deficit that precluded informed consent
* Unwillingness to be followed up for 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-04; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Arthritis of the Shoulder Index (WOOS) | 6 weeks, 3 mo, 6 mo, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr post-op
  The WOOS will be done at 6 weeks, 3 months, 6 months and yearly post-op to compare with the baseline pre-op score.

SECONDARY OUTCOMES:
Change in ASES score | 6 weeks, 3 mo, 6 mo, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr post-op
  The ASES will be done at 6 weeks, 3 months, 6 months and yearly post-op to compare with the baseline pre-op score.
Change in Short Form 12 (SF-12) | 6 weeks, 3 mo, 6 mo, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr post-op
  The SF-12 will be done at 6 weeks, 3 months, 6 months and yearly post-op to compare with the baseline pre-op score.
Change in Health Resource Utilization Instrument | 6 weeks, 3 mo, 6 mo, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr post-op
  The Health Resource Utilization Instrument will be done at 6 weeks, 3 months, 6 months and yearly post-op to gather data on the associated costs of the respective surgeries.
Change in Radiographic evaluation | post-op day 0 or 1, 6 weeks, 3 months, 6 months, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr post-op
  Grashey A-P and axillary views to assess component position, metallic debris, and radiolucency in 6 zones post op.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chin, MD,FRCSC,MBA, Principal Investigator — Joint Preservation Centre of BC/University of British Columbia
Locations (6):
- Canada (6):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Richmond General Hospital, Richmond, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia